CLINICAL TRIAL: NCT04845672
Title: Comparison of the Permanent Skin Flora of Children Who Had Bathing With Two Different Products: A Randomized Controlled Study
Brief Title: Comparison of the Permanent Skin Flora of Children Who Had Bathing With Two Different Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, cagri covener ozcelik, Assoc.Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01/28
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Skin Microbiota
Keywords: Microbiota; Skin Flora; Wipe Bath; Chlorhexidine Gluconate; Soap-Free Body Wash Solution
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% chlorhexidine gluconate (Experimental): 4% Chlorhexidine gluconate solution and one to one water will be used to create a 2% Chlorhexidine gluconate solution.
  Interventions: Other: 2% chlorhexidine gluconate
- soap-free body cleaning solution (Active Comparator): It supports and protects the natural barrier function of the skin's natural protective layer.
  Interventions: Other: soap-free body cleaning solution

INTERVENTIONS:
Other: 2% chlorhexidine gluconate — Children in 2% chlorhexidine gluconate group , which is the routine practice of the hospital, and a wiping bath in accordance with the bath protocol specified. The bath procedure will take 10-15 minutes. Before wiping bath swab sample will provide from armpit and groin with circular manner and 6 hours later swap sample will be provided from the same areas again. The swab sample taken will be planted on blood agar medium and kept at + 4-8 ℃ for an average of 18-24 hours. After it is planted on blood agar medium, it will be kept at + 4-8 ℃ for an average of 18-24 hours . A total of 12 swab samples will be taken for 3 days from each child and from the same areas, body flora will be evaluated.
  Arms: 2% chlorhexidine gluconate
Other: soap-free body cleaning solution — Children in a wiping bath with soap-free body washing solution group, and a wiping bath in accordance with the bath protocol specified. The bath procedure will take 10-15 minutes. Before wiping bath swab sample will provide from armpit and groin with circular manner and 6 hours later swap sample will be provided from the same areas again. The swab sample taken will be planted on blood agar medium and kept at + 4-8 ℃ for an average of 18-24 hours. After it is planted on blood agar medium, it will be kept at + 4-8 ℃ for an average of 18-24 hours . A total of 12 swab samples will be taken for 3 days from each child and from the same areas, body flora will be evaluated.
  Arms: soap-free body cleaning solution

SUMMARY:
This study was carried out as a randomized controlled experimental study to compare the effect of wiping bath with 2% daily chlorhexidine gluconate and soap-free body wash on the permanent skin flora of children hospitalized in the PICU.

DETAILED DESCRIPTION:
Microbiota to the ecosystem formed by symbiotic and pathogenic microorganisms (bacteria, fungi, viruses, archaea, etc.) living in and on the surface of the human body; All of the genes encoding them have been called the microbiome (Whitman et al., 1998). The relationship between microbiota and many diseases that will have important consequences in human life has been proven. Infection and infectious diseases increase the risk of developing complications in critically ill patients, sometimes followed by death. Microbiota in healthy individuals contains many different microorganisms. The microbiota that begins to form immediately after birth varies according to nutrition, genetics, age and geographic region and climate. Human microbiota may change after applications such as infections, use of antibiotics, various chemicals (antiseptic solutions, soaps, shampoos, etc.). This study was planned to compare the effect of wiping bath with 2% daily chlorhexidine gluconate and soap-free body washing solution on the skin microbiota of the patients hospitalized in the PICU. This research will be done as a randomized controlled experimental. The research population consists of 30 pediatric patients hospitalized in the Pediatric Intensive Care Unit of the Health Sciences University Umraniye Training and Research Hospital in 2021, who were wiped with 2% chlorhexidine gluconate, and 30 who were wiped with a soap-free body wash solution. Power analysis was erformed using the G * Power (v3.1.7) program to determine the number of samples. The strength of the study is expressed as 1-β (= type II error probability) and generally the studies should have 80% power. According to Cohen's effect size coefficients; Assuming that the evaluations to be made between two independent groups will have a large effect size (d = 0.8), it was decided to recruit 30 people, considering that there should be at least 26 people in each group at the level of α = 0.05 and there might be losses in the working process. The research sample was randomly divided into branches; group I will consist of 30 patients and group II will consist of 30 patients. Children in Group I will be applied soap-free body washing solution and children in Group II will be applied a wipe bath with 2% chlorhexidinegluconate, which is the routine application of the unit. In both groups, swab samples will be taken from the right armpit and right groin before and after the wipe bath (6th hour). '' Child Identification Form'' and ''Wipe Bathroom Application Chart'' will be used to collect data. The Child Diagnostic Form consists of questions containing information about the child (age, gender, reason for hospitalization, date, etc.). It is planned to record information on the wiping bath application schedule, the skin reactions that may occur in the patient during the wiping bath and the effect on the skin flora in the swab samples taken before and after the children's bath applications. Data collection tools will be filled in by the researcher through observation. During the data collection process, it was decided by the researcher to take swab samples before each wipe bath application and after the wipe bath application (6th hour) in order to check whether there was growth in the skin flora of the child's armpit and groin areas. Before the research, the parents of the participants will be informed about the research and verbal / written consent will be obtained from the parents declaring their acceptance to participate in the study. Collected data will be evaluated using the SPSS Statistics 22 package program. At the end of the study, it is thought that it will guide the improvement of patient care quality.

ELIGIBILITY:
Inclusion Criteria:

* Being in the first 24 hours of admission to the PICU
* Internal reasons for hospitalization with children
* No co-morbid disease
* Hospitalization in PICU during data collection procedure

Exclusion Criteria:

* Hospitalization just before the study
* The children who is not available for wiping bath
* Hospitalized children after surgical procedures
* Antibotic use during the study
* Being chlorhexidine gluconate allergy history
* Impaired skin integrity (burns, skin disease etc.)
* Use of antibiotics, probiotics or steroid-containing immune system suppressing agents at last two months
* Radiotherapy or the chemotherapy patients
* Severe septic shock
* The children with tracheostomy, PEG, permanent dialysis catheter etc.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
permanent skin flora | 3 days
  Blood Agar Base will be used to evaluate permanent skin flora

CONTACTS AND LOCATIONS:
Locations (1):
- Çağrı Çövener Özçelik, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow J, Lee SM, Shen Y, Khosravi A, Mazmanian SK. Host-bacterial symbiosis in health and disease. Adv Immunol. 2010;107:243-74. doi: 10.1016/B978-0-12-381300-8.00008-3. PMID 21034976
- [Background] Clemente JC, Ursell LK, Parfrey LW, Knight R. The impact of the gut microbiota on human health: an integrative view. Cell. 2012 Mar 16;148(6):1258-70. doi: 10.1016/j.cell.2012.01.035. PMID 22424233
- [Background] Costello EK, Lauber CL, Hamady M, Fierer N, Gordon JI, Knight R. Bacterial community variation in human body habitats across space and time. Science. 2009 Dec 18;326(5960):1694-7. doi: 10.1126/science.1177486. Epub 2009 Nov 5. PMID 19892944
- [Background] Elias PM. Stratum corneum defensive functions: an integrated view. J Invest Dermatol. 2005 Aug;125(2):183-200. doi: 10.1111/j.0022-202X.2005.23668.x. PMID 16098026
- [Background] Human Microbiome Project Consortium. A framework for human microbiome research. Nature. 2012 Jun 13;486(7402):215-21. doi: 10.1038/nature11209. PMID 22699610
- [Result] Karki S, Cheng AC. Impact of non-rinse skin cleansing with chlorhexidine gluconate on prevention of healthcare-associated infections and colonization with multi-resistant organisms: a systematic review. J Hosp Infect. 2012 Oct;82(2):71-84. doi: 10.1016/j.jhin.2012.07.005. Epub 2012 Aug 11. PMID 22889522
- [Result] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Result] Kong HH, Segre JA. Skin microbiome: looking back to move forward. J Invest Dermatol. 2012 Mar;132(3 Pt 2):933-9. doi: 10.1038/jid.2011.417. Epub 2011 Dec 22. PMID 22189793
- [Result] Whitman WB, Coleman DC, Wiebe WJ. Prokaryotes: the unseen majority. Proc Natl Acad Sci U S A. 1998 Jun 9;95(12):6578-83. doi: 10.1073/pnas.95.12.6578. PMID 9618454